CLINICAL TRIAL: NCT07139912
Title: Prospective, Multicenter, Single-Arm Trial Assessing Safety/Effectiveness of Multi-Branch Thoracic Stent Grafts in Aortic Arch Disease
Brief Title: Prospective, Multicenter, Single-Arm Study of Aortic Arch Pathology Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Endovascular MedTech（Group）Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endovastec
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Aortic Arch Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group/Arm (Experimental): Participants will be treated with Thoracic Aortic Multi-Branch Stent Graft System, developed and manufactured by Shanghai MicroPort Endovascular MedTech (Group) Co., Ltd
  Interventions: Device: Thoracic Aortic Multi-Branch Stent Graft System

INTERVENTIONS:
Device: Thoracic Aortic Multi-Branch Stent Graft System — The Thoracic Aortic Multi-Branch Stent Graft Systemm consists of the Single-Branch Aortic Stent-Graft System, the aortic extension stent graft system and the branch stent system.

SUMMARY:
A prospective ,multiple center Study about the Safety and Efficacy of the Thoracic Aortic Multi-Branch Stent Graft System, developed and manufactured by Shanghai MicroPort Endovascular MedTech (Group) Co., Ltd., in patients with aortic arch pathologies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years
2. Diagnosed with aortic arch pathology requiring intervention, including:

   True aortic arch aneurysm

   Pseudoaneurysm of the aortic arch

   Penetrating aortic ulcer involving the arch
3. Deemed suitable for endovascular repair by the investigating physician
4. Capable of understanding study objectives, providing written informed consent, and complying with follow-up requirements
5. Anatomic suitability confirmed by CTA:

   Ascending aortic length ≥50 mm

   Ascending aortic diameter ≥26 mm and ≤46 mm

   Proximal landing zone length ≥20 mm

   Brachiocephalic trunk diameter ≥9 mm and ≤19 mm with length ≥20 mm

   Left common carotid artery (LCCA) and left subclavian artery (LSA) diameters ≥5 mm and ≤13 mm

   LCCA length ≥20 mm

   Distance from LSA ostium to left vertebral artery origin ≥20 mm
6. High surgical risk per investigator assessment OR contraindicated for open surgery

Exclusion Criteria:

1. Pregnant or lactating women
2. Connective tissue disorders affecting the aorta (e.g., Marfan syndrome, Ehlers-Danlos syndrome)
3. Infected aortic pathologies or aortitis (e.g., mycotic aneurysm, Takayasu arteritis)
4. Prior endovascular repair of ascending aorta/aortic arch
5. Documented allergy to nitinol, contrast media, or device materials
6. Severe renal impairment:(Serum creatinine >2×ULN,Excluding dialysis-dependent patients)
7. Hematologic abnormalities:(WBC <3×10⁹/L、Hb <70 g/L、PLT <50×10⁹/L)
8. Heart transplant recipients
9. Myocardial infarction or stroke within 3 months
10. NYHA Class IV heart failure
11. Active systemic infection (e.g., bacteremia, sepsis)
12. Life expectancy <12 months
13. Mechanical aortic valve prosthesis impeding device delivery
14. Current participation in other interventional trials with primary endpoint pending
15. Anticipated poor compliance with follow-up
16. Other contraindications for endovascular repair per investigator assessment:Severe vascular stenosis/calcification/tortuosity/Thrombus at landing zones/Inability to cooperate with procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
12-month treatment success rate | 12-month
  Technical success at the index procedure, without device- or aortic pathology-related mortality or unplanned secondary interventions, and with no evidence of persistent enlargement of the treated aortic segment due to Type I/III endoleaks on 12-month CTA follow-up.
30-day rate of Major Adverse Events (MAE) | 30-day
  Including all-cause mortality, disabling stroke, persistent paraplegia, renal failure, myocardial infarction, and respiratory failure

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No